CLINICAL TRIAL: NCT00067119
Title: Effect of Dipyridamole Plus Aspirin on Hemodialysis Graft Patency
Brief Title: Aggrenox Prevention of Access Stenosis
Acronym: GRAFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The Cleveland Clinic (Other); Boston University (Other); Duke University (Other); University of Iowa (Other); MaineHealth (Other); University of Texas Southwestern Medical Center (Other); University of Alabama at Birmingham (Other); Washington University School of Medicine (Other); Baystate Medical Center (Other); Vanderbilt University (Other); CAMC Health System (Other); Emory University (Other); St. Louis University (Other); Tyler Nephrology Associates (Unknown); Vascular Surgery Associates LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC GRAFT; U01DK058982 (NIH)
Record Dates: First submitted 2003-08-11; First posted 2003-08-13 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Kidney Failure
Keywords: Graft Failure; Access Blood Flow Monitoring; Clinical Trial Vascular Access; Fistula Failure; Hemodialysis; Vascular Access
MeSH Terms: conditions — Renal Insufficiency | interventions — Aspirin, Dipyridamole Drug Combination; Dipyridamole; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aggrenox (Experimental)
  Interventions: Drug: Aggrenox
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aggrenox
  Other Names: Dipyridamole plus aspirin
  Arms: Aggrenox
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to determine whether Aggrenox (Boehringer-Ingelheim) prolongs primary unassisted patency in newly created arteriovenous grafts. This record previously included information for both the GRAFT and FISTULA trials.

ELIGIBILITY:
Inclusion criteria:

* Age 18-21 depending on state regulations
* Life expectancy of at least six months
* Chronic renal failure with anticipated start of hemodialysis within six months of enrollment, or current dialysis dependence
* A new or planned arteriovenous (AV) graft placed in any location for the purpose of hemodialysis. (Any type of graft material and any configuration of the access is acceptable).
* The patient is expected to stay at a participating dialysis facility for at least 6 months.
* The patient's physician(s) will allow the patient to participate.
* Ability to give informed consent.

Exclusion Criteria:

* Women must not be pregnant, breastfeeding, or plan to be pregnant during the course of the study.
* The presence of ongoing bleeding.
* The presence of a known bleeding disorder (e.g., hemophilia or von Willebrand's disease).
* Recent bleeding episode requiring transfusion within 12 weeks of entry.
* The presence of acute ulcer disease. Acute ulcer disease is defined as a new diagnosis of peptic disease including esophagitis, gastritis, or ulcer or the initiation of treatment with proton pump inhibitors, H2 blockers or therapy for Helicobacter pylori within three months prior to obtaining consent.
* Known allergy or adverse reaction to Aggrenox or any of its study components (dipyridamole and aspirin).
* Required use of warfarin, dipyridamole, non-steroidal antiinflammatory drugs or other antiplatelet agents other than aspirin.
* Current uncontrolled hypertension with systolic blood pressure in excess of 200 mm Hg or diastolic blood pressure in excess of 115 mm Hg.
* Baseline platelet count less than 75,000/mm3.
* Known advanced liver disease with decompensated cirrhosis, jaundice, ascites or bleeding varices.
* Current problem with substance abuse.
* Concurrent participation in another medical intervention trial.
* Anticipated non-compliance with medical care based on physician judgment.
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2008-01-31 (Actual); Study Completion 2008-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Kusek, Ph.D., Study Director — NIDDK - Telephone: 301-594-7717; Email: kusekj@ep.niddk.nih.gov; Catherine Meyers, M.D., Study Director — NIDDK - Telephone: 301-451-4901; Email: meyersc@extra.niddk.nih.gov
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Iowa, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Boston University Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the National Institute of Diabetes Digestive and Kidney Diseases (NIDDK) Central Repository
Time Frame: Data were available in December 2011
URL: https://www.niddkrepository.org/studies/graft/?query=dac

REFERENCES:
- [Background] Dixon BS, Beck GJ, Dember LM, Depner TA, Gassman JJ, Greene T, Himmelfarb J, Hunsicker LG, Kaufman JS, Lawson JH, Meyers CM, Middleton JP, Radeva M, Schwab SJ, Whiting JF, Feldman HI; DAC Study Group. Design of the Dialysis Access Consortium (DAC) Aggrenox Prevention Of Access Stenosis Trial. Clin Trials. 2005;2(5):400-12. doi: 10.1191/1740774505cn110oa. PMID 16317809
- [Result] Dixon BS, Beck GJ, Vazquez MA, Greenberg A, Delmez JA, Allon M, Dember LM, Himmelfarb J, Gassman JJ, Greene T, Radeva MK, Davidson IJ, Ikizler TA, Braden GL, Fenves AZ, Kaufman JS, Cotton JR Jr, Martin KJ, McNeil JW, Rahman A, Lawson JH, Whiting JF, Hu B, Meyers CM, Kusek JW, Feldman HI; DAC Study Group. Effect of dipyridamole plus aspirin on hemodialysis graft patency. N Engl J Med. 2009 May 21;360(21):2191-201. doi: 10.1056/NEJMoa0805840. PMID 19458364
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Mohamed I, Kamarizan MFA, Da Silva A. Medical adjuvant treatment to increase patency of arteriovenous fistulae and grafts. Cochrane Database Syst Rev. 2021 Jul 23;7(7):CD002786. doi: 10.1002/14651858.CD002786.pub4. PMID 34298589
- [Derived] Dember LM, Beck GJ, Allon M, Delmez JA, Dixon BS, Greenberg A, Himmelfarb J, Vazquez MA, Gassman JJ, Greene T, Radeva MK, Braden GL, Ikizler TA, Rocco MV, Davidson IJ, Kaufman JS, Meyers CM, Kusek JW, Feldman HI; Dialysis Access Consortium Study Group. Effect of clopidogrel on early failure of arteriovenous fistulas for hemodialysis: a randomized controlled trial. JAMA. 2008 May 14;299(18):2164-71. doi: 10.1001/jama.299.18.2164. PMID 18477783